CLINICAL TRIAL: NCT01844765
Title: A Multi-center, Open Label, Non-controlled Phase II Study to Evaluate Efficacy and Safety of Oral Nilotinib in Pediatric Patients With Newly Diagnosed Ph+ Chronic Myelogenous Leukemia (CML) in Chronic Phase (CP) or With Ph+ CML in CP or Accelerated Phase (AP) Resistant or Intolerant to Either Imatinib or Dasatinib
Brief Title: Open Label, Phase II Study to Evaluate Efficacy and Safety of Oral Nilotinib in Philadelphia Positive (Ph+) Chronic Myelogenous Leukemia (CML) Pediatric Patients.
Acronym: DIALOG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107A2203; 2013-000200-41 (EudraCT Number)
Expanded Access: NCT04518644 (No longer available)
Record Dates: First submitted 2013-04-29; First posted 2013-05-01 (Estimated); Results first posted 2018-05-21 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-03

CONDITIONS: Philadelphia Positive (Ph+) Chronic Myelogenous Leukemia
Keywords: Tasigna; nilotinib treatment; chronic phase; Ph+ CML; accelerated phase; newly diagnosed Ph+ CML; pediatric; leukemia; leukemia, pediatric; leukemia, myleiod; leukemia, mylegenous, chronic; leukemia, mylegenous, accelerated; BCR-ABL positive; myeloproliferative disorder; bone marrow disease; hematologic diseases; neoplastic processes; imatinib; dasatinib; enzyme inhibitor; protein kinase inhibitor
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia; Bronchiolitis Obliterans Syndrome; Myeloproliferative Disorders; Bone Marrow Diseases; Hematologic Diseases; Neoplastic Processes | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Newly diagnosed and untreated Ph+ CML in first CP (Experimental): Diagnosis within 6 months of date of first cytogenetic analysis confirming Philadelphia chromosome with (9;22) translocation by standard conventional cytogenetic analysis.
  Interventions: Drug: nilotinib
- Resistant/intolerant Ph+ CML in CP (Experimental): Resistant or Intolerant to either imatinib or dasatinib
  Interventions: Drug: nilotinib
- Resistant/intolerant Ph+ CML in AP (Experimental): Resistant or intolerant to either imatinib or dasatinib - at the end no patients were enrolled in this arm.
  Interventions: Drug: nilotinib

INTERVENTIONS:
Drug: nilotinib — Nilotinib supplied in 50mg, 150mg, and 200mg capsules. It was administered orally at 230mg/m2, twice daily for up to 66 cycles (1 cycle = 28 days). Dose administration was rounded to the nearest 50mg dose (to a maximum dose of 400mg).
  Other Names: AMN107

SUMMARY:
To evaluate the safety, efficacy and pharmacokinetics of nilotinib over time in the Ph+ chronic myelogenous leukemia (CML) in pediatric patients (from 1 to <18 years).

DETAILED DESCRIPTION:
The study was designed as a multi-center, open-label, non-controlled phase II study to assess efficacy, safety and PK parameters of 230 mg/m2 twice daily nilotinib in pediatric patients (1 to <18 years old). The study population consisted of three cohorts of Ph+ CML pediatric patients:

* Cohort 1: Ph+ CML-CP patients resistant or intolerant to either imatinib or dasatinib
* Cohort 2: Ph+ CML-AP patients resistant or intolerant to either imatinib or dasatinib
* Cohort 3: Newly-diagnosed Ph+ CML-CP patients in first chronic phase A minimum number of 50 pediatric patients (from 1 to <18 years) were enrolled in the study. Of them, at least 15 patients were Ph+ CML-CP patients resistant or intolerant to either imatinib or dasatinib, and at least 15 were newly-diagnosed Ph+ CML-CP patients in first chronic phase patients. There was no minimum number of patients required for Ph+ CML-AP patients resistant or intolerant to either imatinib or dasatinib.

Based on enrollment forecasts as of Jan 2015, and to reflect the agreements with the US FDA and the PDCO, the study remained open for enrollment until the targeted number of 50 patients with at least 15 newly diagnosed Ph+CML patients was achieved or until 31May2015, whichever was later.

Patients who completed the study were treated with nilotinib for a total of 66 cycles of 28 days unless the patient prematurely discontinued study treatment.

The primary analysis cut-off date was the date when all patients enrolled in the trial either completed their visit for treatment cycle 12 or had discontinued study treatment early (EoT/early discontinuation visit). These analyses were reported in the 12-cycle clinical study report (CSR). A 24-cycle analysis was done when all patients had either completed their 24-cycle treatment visit or had discontinued study treatment early.

At trial end, a final comprehensive CSR of all data collected during the trial was produced.

ELIGIBILITY:
Key Inclusion Criteria:

* Newly diagnosed and untreated Ph+ CML CP or Ph+ CML CP or AP resistant or intolerant to either imatinib or dasatinib
* Karnofsky ≥ 50% for patients > 10 years of age and Lansky ≥ 50 for patients ≤ 10 years of age
* Adequate renal, hepatic and pancreatic function
* Potassium, magnesium, phosphorus and total calcium values ≥ LLN (lower limit of normal)
* Written informed consent

Key Exclusion Criteria:

* Treatment with strong CYP3A4 inhibitors or inducers
* Use or planned use of any medications that have a known risk or possible risk to prolong the QT interval
* Acute or chronic liver, pancreatic or severe renal disease
* History of pancreatitis or chronic pancreatitis.
* Impaired cardiac function
* No evidence of active graft vs host and <3mo since Stem Cell Transplant
* Total body irradiation (TBI) or craniospinal radiation therapy <6months
* Hypersensitivity to the active ingredient or any of the excipients including lactose.
* the criteria regarding pregnancy and contraception
* Active or systemic bacterial, fungal, or viral infection
* known Hepatitis B, Hepatitis C, or HIV infection

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2013-08-20 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2020-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (34):
- United States (10):
  - Loma Linda University Cancer Center, Loma Linda, California
  - Lucile Salter Packard Children's Hospital at Stanford, Palo Alto, California
  - Nemours Childrens Hospital, Orlando, Florida
  - St. Mary's Hospital, West Palm Beach, Florida
  - Johns Hopkins Oncology Center ORA, Baltimore, Maryland
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - Nationwide Childrens Hospital, Columbus, Ohio
  - University of Texas Southwestern Medical Center Oncology, Dallas, Texas
  - Cook Children's Medical Center Oncology, Fort Worth, Texas
  - Seattle Childrens Hospital, Seattle, Washington
- France (4):
  - Novartis Investigative Site, Bordeaux, Aquitaine
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Poitiers
- Novartis Investigative Site, Budapest, Hungary
- Italy (4):
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Torino, TO
- Japan (5):
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Sakyo Ku, Kyoto
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Saitama
  - Novartis Investigative Site, Shizuoka
- Novartis Investigative Site, Kuala Lumpur, Malaysia
- Novartis Investigative Site, Rotterdam, Netherlands
- Novartis Investigative Site, Moscow, Russia
- Novartis Investigative Site, Seoul, South Korea
- Novartis Investigative Site, Madrid, Spain
- Thailand (2):
  - Novartis Investigative Site, Muang, Chiangmai
  - Novartis Investigative Site, Bangkok
- Novartis Investigative Site, Istanbul, Turkey (Türkiye)
- United Kingdom (2):
  - Novartis Investigative Site, Sutton, Surrey
  - Novartis Investigative Site, Bristol

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Hijiya N, Maschan A, Rizzari C, Shimada H, Dufour C, Goto H, Kang HJ, Guinipero T, Karakas Z, Bautista F, Ducassou S, Yoo KH, Zwaan CM, Millot F, Patterson BC, Samis J, Izquierdo M, Titorenko K, Li S, Sosothikul D. The long-term efficacy and safety of nilotinib in pediatric patients with CML: a 5-year update of the DIALOG study. Blood Adv. 2023 Dec 12;7(23):7279-7289. doi: 10.1182/bloodadvances.2023010122. PMID 37738125
- [Derived] Hijiya N, Maschan A, Rizzari C, Shimada H, Dufour C, Goto H, Kang HJ, Guinipero T, Karakas Z, Bautista F, Ducassou S, Yoo KH, Zwaan CM, Millot F, Patterson B, Samis J, Aimone P, Allepuz A, Titorenko K, Sosothikul D. A phase 2 study of nilotinib in pediatric patients with CML: long-term update on growth retardation and safety. Blood Adv. 2021 Jul 27;5(14):2925-2934. doi: 10.1182/bloodadvances.2020003759. PMID 34309636
- [Derived] Hijiya N, Maschan A, Rizzari C, Shimada H, Dufour C, Goto H, Kang HJ, Guinipero T, Karakas Z, Bautista F, Ducassou S, Yoo KH, Zwaan CM, Millot F, Aimone P, Allepuz A, Quenet S, Hourcade-Potelleret F, Hertle S, Sosothikul D. Phase 2 study of nilotinib in pediatric patients with Philadelphia chromosome-positive chronic myeloid leukemia. Blood. 2019 Dec 5;134(23):2036-2045. doi: 10.1182/blood.2019000069. PMID 31511239

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3 cohorts were planned based on disease classification. In 1 cohort no patients (pts) were enrolled so results presented are based on 2 cohorts. 34 imatinib/dasatinib resistant/intolerant CML-CP pts & 25 newly diagnosed CML-CP pts were enrolled. 1 imatinib/dasatinib resistant/intolerant pt did not receive study drug & was excluded from analysis.
Pre-assignment Details: Minimum 50 pediatric patients (pts) to be enrolled in the study. At least 15 were to be Ph+ CML-CP pts resistant/intolerant to either imatinib or dasatinib, & at least 15 newly diagnosed Ph+ CML-CP pts. There was no requirement on the minimum number of pts to be enrolled in the Cohort of CML-AP resistant/intolerant to either imatinib or dasatinib.
Groups:
- Resistant/Intolerant Ph+ CML in CP: Patients resistant or intolerant to either imatinib or dasatinib
- Newly Diagnosed and Untreated Ph+ CML in First CP: Patients newly diagnosed in Chronic phase. Diagnosis within 6 months of date of first cytogenetic analysis confirming Philadelphia chromosome with (9;22) translocation by standard conventional cytogenetic analysis
Period: Overall Study
Arm/Group | Resistant/Intolerant Ph+ CML in CP | Newly Diagnosed and Untreated Ph+ CML in First CP
Started | 34 | 25
Treated | 33 | 25
Untreated | 1 (Did not receive study drug due to adverse event (AE).) | 0
Completed (Completed = Treatment duration is completed per protocol) | 19 | 10
Not Completed | 15 | 15
Not completed — Adverse Event | 6 | 8
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Disease progression | 1 | 0
Not completed — Administrative problems | 3 | 4
Not completed — Protocol deviation | 2 | 0
Not completed — Untreated | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All patients who received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Resistant/Intolerant Ph+ CML in CP | Newly Diagnosed and Untreated Ph+ CML in First CP | Total
Number analyzed (Participants) | 33 | 25 | 58
Age, Customized [Number; unit: Participants] — Population: Full Analysis Set (FAS): All patients who received at least one dose of study medication.
  Participants
    1 to < 12 years | 12 | 6 | 18
    12 to < 18 years | 21 | 19 | 40
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Full Analysis Set (FAS): All patients who received at least one dose of study medication.
  Participants
    Female | 12 | 12 | 24
    Male | 21 | 13 | 34
Race/Ethnicity, Customized [Number; unit: Participants] — Population: Full Analysis Set (FAS): All patients who received at least one dose of study medication.
  Participants
    Caucasian | 12 | 18 | 30
    Black | 3 | 0 | 3
    Asian | 16 | 7 | 23
    Native American | 1 | 0 | 1
    Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Rate of Major Molecular Response (MMR) at 6 Cycles for Ph+ CML CP Patients Resistant or Intolerant to Imatinib or Dasatinib
Description: MMR is defined as ≤ 0.1% BCR-ABL/control gene (ABL) % by international scale, or equivalent to ≥ 3 log reduction of BCR-ABL transcript from standardized baseline, measured by RQ-PCR (Real time quantitative polymerase chain reaction). BCR-ABL is the fusion gene from breakpoint cluster region and Abelson genes. A patient was counted as having MMR at 6 cycles if the patient met the MMR criteria at the Cycle 6 Visit.
Time Frame: 6 cycles
Population: Full Analysis Set (FAS): All patients who received at least one dose of study medication
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Resistant/Intolerant Ph+ CML in CP
Number analyzed (Participants) | 33
Percentage of participants | 39.4 [22.9 to 57.9]

2. Primary Outcome: MMR Rate by 12 Cycles in Newly Diagnosed Ph+ CML-CP Patients
Description: MMR is defined as ≤ 0.1% BCR-ABL/control gene (ABL) % by international scale, or equivalent to ≥ 3 log reduction of BCR-ABL transcript from standardized baseline, measured by RQ-PCR (Real time quantitative polymerase chain reaction). BCR-ABL is the fusion gene from breakpoint cluster region and Abelson genes. A patient was counted as having MMR by 12 cycles if the patient met the MMR criteria at least once at any time between first study drug intake and Cycle 12 visit included.
Time Frame: 12 cycles
Population: Full Analysis Set (FAS): All patients who received at least one dose of study medication
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Newly Diagnosed and Untreated Ph+ CML in First CP
Number analyzed (Participants) | 25
Percentage of participants | 64.0 [42.5 to 82.0]

3. Primary Outcome: Rate of Complete Cytogenic Response (CCyR) at 12 Cycles in Newly Diagnosed Ph+ CML-CP Patients
Description: Cytogenetic response is assessed as the percentage of Philadelphia positive (Ph+) metaphases in the bone marrow. Complete Cytogenetic Response (CCyR) is defined as 0% of Ph+ metaphases. A patient was counted as CCyR at 12 cycles if the patient met the CCyR criteria at the Cycle 12 Visit.
Time Frame: 12 cycles
Population: Full Analysis Set (FAS): All patients who received at least one dose of study medication
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Newly Diagnosed and Untreated Ph+ CML in First CP
Number analyzed (Participants) | 25
Percentage of participants | 64.0 [42.5 to 82.0]

4. Secondary Outcome: MMR Rate by Time Points in Ph+ CML-CP Patients Resistant or Intolerant to Imatinib or Dasatinib
Description: Major molecular response (MMR) was defined as BCR-ABL/ABL % ≤ 0.1% by IS as measured by RQ-PCR, confirmed by duplicate analysis of the same sample.
Time Frame: By 3, 6, 9 , 12, 24, 36, 48, 66 cycles ( 1 cycle = 28 days)
Population: Full Analysis Set (FAS): All patients who received at least one dose of study medication
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Resistant/Intolerant Ph+ CML in CP
Number analyzed (Participants) | 33
Percentage of participants
  By cycle 3 | 36.4 [20.4 to 54.9]
  By cycle 6 | 45.5 [28.1 to 63.6]
  By cycle 9 | 51.5 [33.5 to 69.2]
  By cycle 12 | 57.6 [39.2 to 74.5]
  By cycle 18 | 57.6 [39.2 to 74.5]
  By cycle 24 | 57.6 [39.2 to 74.5]
  By cycle 36 | 57.6 [39.2 to 74.5]
  By cycle 48 | 60.6 [42.1 to 77.1]
  By cycle 66 | 60.6 [42.1 to 77.1]

5. Secondary Outcome: MMR Rate by Time Points in Newly Diagnosed Ph+ CML-CP Patients
Description: as for outcome 4
Time Frame: by 3, 6, 9, 12, 24, 36, 48, 66 cycles (1 cycle = 28 days)
Population: Full Analysis Set (FAS): All patients who received at least one dose of study medication
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Newly Diagnosed and Untreated Ph+ CML in First CP
Number analyzed (Participants) | 25
Percentage of participants
  By cycle 3 | 12.0 [2.5 to 31.2]
  By cycle 6 | 52.0 [31.3 to 72.2]
  By cycle 9 | 56.0 [34.9 to 75.6]
  By cycle 12 | 64.0 [42.5 to 82.0]
  By cycle 18 | 68.0 [46.5 to 85.1]
  By cycle 24 | 68.0 [46.5 to 85.1]
  By cycle 36 | 76.0 [54.9 to 90.6]
  By cycle 48 | 76.0 [54.9 to 90.6]
  By cycle 66 | 76.0 [54.9 to 90.6]

6. Secondary Outcome: Best BCR-ABL Ratio Categories for Resistant/Intolerant Ph+ CML - Overall
Description: MMR is defined as ≤ 0.1% BCR-ABL/control gene (ABL) % by international scale, or equivalent to ≥ 3 log reduction of BCR-ABL transcript from standardized baseline, measured by RQ-PCR (Real time quantitative polymerase chain reaction). BCR-ABL is the fusion gene from breakpoint cluster region and Abelson genes. BCR-ABL ratio by percentage: > 0.0032 to ≤ 0.01% is equal to a log reduction category of >= 4 to <4.5 -log reduction (MR4); BCR-ABL ratio by percentage: <=0.0032% is equal to a log reduction category of >= 4.5-log reduction (MMR4.5)
Time Frame: up to 66 cycles (1 cycle = 28 days)
Population: Full Analysis Set (FAS): All patients who received at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Resistant/Intolerant Ph+ CML in CP
Number analyzed (Participants) | 33
Percentage of participants
  <=0.0032% | 12.1
  > 0.0032% - ≤ 0.01% | 15.2
  >0.01% - ≤ 0.1% | 33.3
  >0.1% - ≤ 1% | 21.2
  >1% - ≤ 10% | 9.1
  > 10% | 6.1
  Atypical transcripts at baseline | 3.0

7. Secondary Outcome: Best BCR-ABL Ratio Categories for Newly Diagnosed Ph+ CML-CP - Overall
Description: as for outcome 6
Time Frame: up to 66 cycles (1 cycle = 28 days)
Population: Full Analysis Set (FAS): All patients who received at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Newly Diagnosed and Untreated Ph+ CML in First CP
Number analyzed (Participants) | 25
Percentage of participants
  ≤ 0.0032% | 44.0
  >0.0032% - ≤ 0.01% | 12.0
  >0.01% - ≤ 0.1% | 20.0
  >0.1% - ≤ 1% | 8.0
  >1% - ≤ 10% | 8.0
  >10% | 8.0

8. Secondary Outcome: Time to First MMR Among Imatinib or Dasatinib Resistant or Intolerant CML-CP Patients Who Achieved MMR
Description: Time from first study drug intake to first MMR amongst imatinib or dasatinib resistant or intolerant patients with CML-CP computed only for patients who achieved MMR.
Time Frame: From first dosing to the first MMR within 66 cycles period
Population: Full Analysis Set (FAS): All patients who received at least one dose of study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Resistant/Intolerant Ph+ CML in CP
Number analyzed (Participants) | 20
months | 2.79 [0.03 to 5.75]

9. Secondary Outcome: Time to First MMR Among Newly Diagnosed Ph+ CML-CP Patients Who Achieved MMR
Description: Time to MMR is the time from first study drug intake to first major molecular response computed only for participants who achieved MMR.
Time Frame: From first dosing to the first MMR within 66 cycles period
Population: Full Analysis Set (FAS): All patients who received at least one dose of study medication.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Newly Diagnosed and Untreated Ph+ CML in First CP
Number analyzed (Participants) | 19
Months | 5.59 [5.52 to 10.84]

10. Secondary Outcome: Duration of First MMR Among Patients Who Were Resistant or Intolerant to Either Imatinib or Dasatinib Who Achieved MMR
Description: Duration of MMR is defined as the time between the date of the first MMR and the date of confirmed loss of MMR (i.e. the earliest of confirmed loss of MMR, CML-related death or progression to AP or BC). Participants without loss of MMR were censored at the last molecular assessment date.
Time Frame: from MMR until confirmed loss of MMR (Assessed up to 66 cycles)
Population: Full Analysis Set (FAS): All patients who received at least one dose of study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Resistant/Intolerant Ph+ CML in CP
Number analyzed (Participants) | 20
months | NA [NA to NA] — NA = not estimable as there were not enough events

11. Secondary Outcome: Duration of First MMR Among Newly Diagnosed Patients Who Achieved MMR
Description: as for outcome 10
Time Frame: from MMR until confirmed loss of MMR (Assessed up to 66 cycles)es)
Population: Full Analysis Set (FAS): All patients who received at least one dose of study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Newly Diagnosed and Untreated Ph+ CML in First CP
Number analyzed (Participants) | 19
months | NA [NA to NA] — NA = not estimable as there were not enough events

12. Secondary Outcome: Best Complete Cytogenetic Response (CCyR) Categories in Ph+ CML-CP Patients Resistant or Intolerant to Imatinib or Dasatinib - Overall
Description: * Complete cytogenetic response (CCyR) - 0% Ph+ metaphases
  * Partial cytogenetic response (PCyR) - >0 to 35% Ph+ metaphases
  * Minor cytogenetic response (mCyR) - >35 to 65% Ph+ metaphases
  * Minimal - >65 to 95% Ph+ metaphases
  * None - >95 to 100% Ph+ metaphases
  * Major cytogenetic response (MCyR) - 0 to 35% Ph+ metaphases. A major response combines both complete and partial responses.
Time Frame: up to 66 cycles
Population: Full Analysis Set (FAS): All patients who received at least one dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Resistant/Intolerant Ph+ CML in CP
Number analyzed (Participants) | 33
Percentage of participants
  Major cytogenetic response: Complete | 81.1
  Major cytogenetic response: Partial | 3.0
  Minimal | 3.0
  None | 3.0
  Missing | 9.1

13. Secondary Outcome: Best Complete Cytogenetic Response (CCyR) in Newly Diagnosed Ph+ CML-CP Patients - Overall
Description: Complete cytogenetic response (CCyR) - 0% Ph+ metaphases No response - >95 to 100% Ph+ metaphases
Time Frame: up to 66 cycles
Population: Full Analysis Set (FAS): All patients who received at least one dose of study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Newly Diagnosed and Untreated Ph+ CML in First CP
Number analyzed (Participants) | 25
Percentage of participants | 84.0 [63.9 to 95.5]

14. Secondary Outcome: Summary of Time to First Complete Cytogenic Response (CCyR) in Newly Diagnosed Ph+ CML-CP Patients
Description: Cytogenetic response is assessed as the percentage of Philadelphia positive (Ph+) metaphases in the bone marrow. Complete Cytogenetic Response (CCyR) is defined as 0% of Ph+ metaphases. A patient was counted as having CCyR by 6 cycles (respectively 12 cycles) if the patient met the CCyR criteria at least once at any time between first study drug intake and cycle 6 (cycle 12 respectively) visit included.
Time Frame: From first dosing to the first CCyR up to 66 cycles
Population: Full Analysis Set (FAS): All patients who received at least one dose of study medication
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Newly Diagnosed and Untreated Ph+ CML in First CP
Number analyzed (Participants) | 25
months | 5.55 [5.49 to 5.59]

15. Secondary Outcome: Kaplan-Meier Estimates of Time to First Complete Cytogenic Response (CCyR) in Newly Diagnosed Ph+ CML-CP Patients
Description: as for outcome 14
Time Frame: From first dosing to the first CCyR up to 66 cycles
Population: Full Analysis Set (FAS): All patients who received at least one dose of study medication
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Newly Diagnosed and Untreated Ph+ CML in First CP
Number analyzed (Participants) | 25
months | 5.6 [5.5 to 5.6]

16. Secondary Outcome: Kaplan-Meier Estimates of Duration of First Complete Cytogenic Response (CCyR) Among Patients Who Achieved CCyR in Newly Diagnosed Ph+ CML-CP Patients
Description: as for outcome 14
Time Frame: From CCyR to loss of CCyR up to 66 cycles
Population: Full Analysis Set (FAS): All patients who received at least one dose of study medication
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Newly Diagnosed and Untreated Ph+ CML in First CP
Number analyzed (Participants) | 21
months | NA [NA to NA] — NA = not estimable as there were not enough events

17. Secondary Outcome: Best Major Cytogenetic Response (MCyR) Rate by Time Point in Newly Diagnosed Ph+ CML Patients
Description: Major cytogenetic response (MCyR) - 0 to 35% Ph+ metaphases. A major response combines both complete and partial responses.
Time Frame: 6, 12, 18, 24, 36, 48, 66 cycles
Population: Full Analysis Set (FAS): All patients who received at least one dose of study medication
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Newly Diagnosed and Untreated Ph+ CML in First CP
Number analyzed (Participants) | 25
Percentage of participants
  by cycle 6 | 88.0 [68.8 to 97.5]
  by cycle 12 | 88.0 [68.8 to 97.5]
  by cycle 18 | 88.0 [68.8 to 97.5]
  by cycle 24 | 88.0 [68.8 to 97.5]
  by cycle 36 | 88.0 [68.8 to 97.5]
  by cycle 48 | 88.0 [68.8 to 97.5]
  by cycle 66 | 88.0 [68.8 to 97.5]

18. Secondary Outcome: Summary of Time to First Major Cytogenetic Response (MCyR) Among Patients Who Achieved MCyR in Newly Diagnosed CML-CP Patients
Description: as for outcome 17
Time Frame: up to 66 cycles
Population: Full Analysis Set (FAS): All patients who received at least one dose of study medication
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Newly Diagnosed and Untreated Ph+ CML in First CP
Number analyzed (Participants) | 22
months | 5.55 [5.52 to 5.59]

19. Secondary Outcome: Kaplan-Meier Estimates of Time to First Major Cytogenetic Response (MCyR) in Newly Diagnosed CML-CP Patients
Description: as for outcome 17
Time Frame: up to 66 cycles
Population: Full Analysis Set (FAS): All patients who received at least one dose of study medication
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Newly Diagnosed and Untreated Ph+ CML in First CP
Number analyzed (Participants) | 25
months | 5.55 [5.52 to 5.59]

20. Secondary Outcome: Best Complete Hematological Response (CHR) by Time Point
Description: Complete Hematological Response (CHR) was defined as
  * WBC count <10×109/L
  * platelet count <450×109/L
  * basophils <5%
  * no blasts and promyelocytes in peripheral blood
  * myelocytes+metamyelocytes <5% in peripheral blood
  * no evidence of extramedullary disease, including spleen and liver
  * Assessment confirmation after at least 4 weeks for newly diagnosed Ph+ CML-CP
Time Frame: cycle 3, 6, 9, 12, 18, 24, 36, 48, 66
Population: Full Analysis Set (FAS): All patients who received at least one dose of study medication
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Newly Diagnosed and Untreated Ph+ CML in First CP
Number analyzed (Participants) | 25
Percentage of participants
  by cycle 3 | 76.0 [54.9 to 90.6]
  by cycle 6 | 84.0 [63.9 to 95.5]
  by cycle 9 | 88.0 [68.8 to 97.5]
  by cycle 12 | 92.0 [74.0 to 99.0]
  by cycle 18 | 92.0 [74.0 to 99.0]
  by cycle 24 | 92.0 [74.0 to 99.0]
  by cycle 36 | 92.0 [74.0 to 99.0]
  by cycle 48 | 92.0 [74.0 to 99.0]
  by cycle 66 | 92.0 [74.0 to 99.0]

21. Secondary Outcome: Summary of Time to First Complete Hematological Response (CHR) Among Patients Who Achieved Confirmed CHR in Newly Diagnosed CML-CP Patients
Description: as for outcome 20
Time Frame: from first dosing to CHR, UP TO 66 CYCLES
Population: Full Analysis Set (FAS): All patients who received at least one dose of study medication
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Newly Diagnosed and Untreated Ph+ CML in First CP
Number analyzed (Participants) | 23
months | 0.95 [0.72 to 2.76]

22. Secondary Outcome: Kaplan-Meier Estimates of Time to First Complete Hematological Response (CHR) in Newly Diagnosed CML-CP Patients
Description: as for outcome 20
Time Frame: from first dosing to CHR, UP TO 66 CYCLES
Population: Full Analysis Set (FAS): All patients who received at least one dose of study medication
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Newly Diagnosed and Untreated Ph+ CML in First CP
Number analyzed (Participants) | 25
months | 1.0 [1.0 to 2.8]

23. Secondary Outcome: Time to Disease Progression for Imatinib or Dasatinib Resistant or Intolerant CML-CP Patients - Kaplan-Meier Estimates
Description: Time to disease progression is the time from the date of first study drug intake to the date of event defined as the first progression to AP or BC (from CP) or to BC (from AP) or the date of CML-related death occurring on treatment, whichever was earlier.
Time Frame: From first dosing to the disease progression within 66 cycles
Population: Full Analysis Set (FAS): All patients who received at least one dose of study medication
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Resistant/Intolerant Ph+ CML in CP
Number analyzed (Participants) | 33
months | NA [NA to NA] — NA = not estimable as there were not enough events

24. Secondary Outcome: Event Free Survival in Imatinib/Dasatinib Resistant/Intolerant CML-CP Patients
Description: Event Free Survival is defined as the time from the date of first study drug intake to the first occurrence of any of the following loss of CHR, loss of MCyR ( PCyR + CCyR), progression to AP/BC (from CP) or to BC (from AP), or death from any cause. (Including events only during treatment)
Time Frame: From first dosing to the disease progression or death up to 66 cycles
Population: Full Analysis Set (FAS): All patients who received at least one dose of study medication
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Resistant/Intolerant Ph+ CML in CP
Number analyzed (Participants) | 33
months | NA [NA to NA] — NA = not estimable as there were not enough events

25. Secondary Outcome: Event Free Survival in Newly Diagnosed CML-CP Patients
Description: as for outcome 24
Time Frame: From first dosing to the disease progression or death up to 66 cycles
Population: Full Analysis Set (FAS): All patients who received at least one dose of study medication
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Newly Diagnosed and Untreated Ph+ CML in First CP
Number analyzed (Participants) | 25
months | NA [NA to NA] — NA = not estimable as there were not enough events

26. Secondary Outcome: Overall Survival (OS) in Imatinib/Dasatinib Resistant/Intolerant CML-CP - Kaplan-Meier Estimates
Description: Overall survival is defined as the time from the date of first study drug intake to the date of death due to any cause. If a patient is not known to have died, survival will be censored at the date of their last assessment for patients on study and date of last contact for patients in follow-up.
Time Frame: from first dosing to death up to 66 cycles
Population: Full Analysis Set (FAS): All patients who received at least one dose of study medication
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Resistant/Intolerant Ph+ CML in CP
Number analyzed (Participants) | 33
months | NA [NA to NA] — NA = not estimable as there were not enough events

27. Secondary Outcome: Overall Survival (OS) in Newly Diagnosed CML-CP Patients
Description: as for outcome 26
Time Frame: from first dosing to death up to 66 cycles
Population: Full Analysis Set (FAS): All patients who received at least one dose of study medication
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Newly Diagnosed and Untreated Ph+ CML in First CP
Number analyzed (Participants) | 25
months | NA [NA to NA] — NA = not estimable as there were not enough events

28. Secondary Outcome: Pharmacodynamics (BCR-ABL Transcript Levels Determined With Standard Protocols in Peripheral Blood): Best MMR Status by Cycle
Description: BCR-ABL is the fusion gene from breakpoint cluster region and Abelson genes. BCR-ABL transcript levels were summarized by cohort and time point. MMR is defined as ≤ 0.1% BCR-ABL/control gene (ABL) % by international scale, or equivalent to ≥ 3 log reduction of BCR-ABL transcript from standardized baseline, measured by RQ-PCR.
Time Frame: By 3, 6, 9, 12, 18, 24, 36, 48, 66 cycles
Population: Full Analysis Set (FAS): All patients who received at least one dose of study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Resistant/Intolerant Ph+ CML in CP | Newly Diagnosed and Untreated Ph+ CML in First CP
Number analyzed (Participants) | 33 | 25
Percentage of participants
  By Cycle 3 | 36.4 [20.4 to 54.9] | 12.0 [2.5 to 31.2]
  By Cycle 6 | 45.5 [28.1 to 63.6] | 52.0 [31.3 to 72.2]
  By Cycle 9 | 51.5 [33.5 to 69.2] | 56.0 [34.9 to 75.6]
  By Cycle 12 | 57.6 [39.2 to 74.5] | 64.0 [42.5 to 82.0]
  By Cycle 18 | 57.6 [39.2 to 74.5] | 68.0 [46.5 to 85.1]
  By Cycle 24 | 57.6 [39.2 to 74.5] | 68.0 [46.5 to 85.1]
  By Cycle 36 | 57.6 [39.2 to 74.5] | 76.0 [54.9 to 90.6]
  By Cycle 48 | 60.6 [42.1 to 77.1] | 76.0 [54.9 to 90.6]
  By Cycle 66 | 60.6 [42.1 to 77.1] | 76.0 [54.9 to 90.6]

29. Secondary Outcome: Pharmacokinetics (PK): Steady State Concentration of Nilotinib in Imatinib/Dasatinib Resistant/Intolerant CML-CP Patients
Description: PK was analyzed only when all patients has completed 12 cycles on treatment or discontinued the study treatment early.
Time Frame: Cycle 1 Day 8
Population: Pharmacokinetics Analysis Set (PAS): All patients with at least one evaluable PK blood sample. Of the 32 patients included in the PAS, only 30 had evaluable Ctrough.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Resistant/Intolerant Ph+ CML in CP
Number analyzed (Participants) | 30
ng/mL | 1407.89 (41.67)

30. Secondary Outcome: Pharmacokinetics: Steady State Concentration of Nilotinib in Newly Diagnosed CML-CP Patients
Description: PK was analyzed only when all patients has completed 12 cycles of treatment or discontinued the study treatment early.
Time Frame: Cycle 1 Day 8
Population: Pharmacokinetics Analysis Set (PAS): All patients with at least one evaluable PK blood sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Newly Diagnosed and Untreated Ph+ CML in First CP
Number analyzed (Participants) | 25
ng/mL | 1274.30 (46.21)

31. Secondary Outcome: Growth Data: Abnormal Height Standard Deviation Scores (SDS) Changes by Cohort
Description: To assess long term effect on growth, development and maturation of nilotinib treatment in pediatric patients with Ph+ CML in participants with both a baseline and post-baseline value.
Time Frame: from first dosing to 66 cycles
Population: Safety Set (SAF): All patients who received at least one dose of study medication in participants with both a baseline and post-baseline value.
Measure: Number; unit: Percentage of participants
Arm/Group | Resistant/Intolerant Ph+ CML in CP | Newly Diagnosed and Untreated Ph+ CML in First CP
Number analyzed (Participants) | 33 | 25
Percentage of participants
  Decrease from baseline of 1 SDS category (n=32,24): number analyzed (Participants) | 32 | 24
  Decrease from baseline of 1 SDS category (n=32,24) | 27.3 | 32.0
  Decrease from baseline of 2 SDS categories (n=32, 24): number analyzed (Participants) | 32 | 24
  Decrease from baseline of 2 SDS categories (n=32, 24) | 3.0 | 16.0
  Decrease from baseline of 3 SDS categories(n= 32, 24): number analyzed (Participants) | 32 | 24
  Decrease from baseline of 3 SDS categories(n= 32, 24) | 6.1 | 4.0

32. Secondary Outcome: Acceptability (Including Palatability) of Dose Forms Used After First Dose, Cycle 1 and Cycle 12 Study Drug Formulation
Description: Acceptability of the study drug was evaluated from a questionnaire completed by patients, with the help from parents or caregivers at visits.
  The Questionnaire to capture patient assessment of palatability (very good to very bad) and acceptability of taking the medication (very easy to very hard to administration).
Time Frame: up to Cycle 12
Population: Safety Set (SAF): All patients who received at least one dose of study medication.
Measure: Number; unit: Percentage of participants
Groups:
- All Patients: All patients enrolled in the study
Arm/Group | All Patients
Number analyzed (Participants) | 58
Percentage of participants
  Cycle (C) 1 Day (D) 1: Completed questionnaire - Patients | 75.9
  C1D1: Completed questionnaire - Parents/Caregivers | 22.4
  C1D1: Patients who swallowed capsule whole | 91.4
  C1D1: Patients had capsule mixed with apple sauce | 6.9
  C1D1: Patients who reported no taste/unable to answer question | 43.1
  C1D1: Patients who reported taste as good/very good | 12.1
  C1D1: Patients who reported taste as not good/not bad | 34.5
  C1D1: Reported capsule to be very easy/easy to administer | 79.3
  C1D28: Completed questionnaire - Patients | 55.2
  C1D28: Completed questionnaire - Parents/Caregivers | 22.4
  C12D28: Completed questionnaire - Patients | 55.2
  C12D28: Completed questionnaire - Parents/Caregivers | 22.4

33. Secondary Outcome: Mutational Assessment of BCR-ABL
Description: Emerging signs of resistance to nilotinib
Time Frame: up to 66 cycles
Population: Full Analysis Set (FAS): All patients who received at least one dose of study medication
Measure: Number; unit: Percentage of participants
Groups:
- Resistant/i Ntolerant Ph+ CML in CP: Patients resistant or intolerant to either imatinib or dasatinib
Arm/Group | Resistant/i Ntolerant Ph+ CML in CP | Newly Diagnosed and Untreated Ph+ CML in First CP
Number analyzed (Participants) | 33 | 25
Percentage of participants
  Patients with >=1 evaluable post-baseline mutational analysis | 39.4 | 32.0
  Patients with any emergent mutation on treatment | 0.0 | 0.0
  Patients with multiple emergent mutations on treatment | 0.0 | 0.0

34. Other Pre Specified Outcome: Long Term Effect of Nilotinib on Bone Metabolism
Description: The summary of bone age and Dual-energy X-ray absorptiometry (DEXA) by cohort. Alteration of bone biochemical markers of hand and wrist X-Ray evaluation was observed in bone age standard deviation scores (SDS) and for bone mineral density for DEXA before and after treatment with nilotinib.
Time Frame: Cycle 66
Population: Safety Set (SAF): All patients who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Percentage of participants
Arm/Group | Resistant/Intolerant Ph+ CML in CP | Newly Diagnosed and Untreated Ph+ CML in First CP
Number analyzed (Participants) | 33 | 25
Percentage of participants
  X-ray (n= 6, 0): number analyzed (Participants) | 6 | 0
  X-ray (n= 6, 0) | -0.61 (1.703) |
  DEXA (n = 14, 10): number analyzed (Participants) | 14 | 10
  DEXA (n = 14, 10) | -0.35 (1.243) | -0.70 (1.043)

35. Post Hoc Outcome: All Collected Deaths
Description: On treatment deaths were collected from FPFT up to 30 days after study drug discontinuation, for a maximum duration of 64.5 months (treatment duration ranged from 0.7 to 63.5 months).
  Deaths post treatment survival follow up were collected after the on- treatment period, up to approx. 7 years.
Time Frame: approx. 64.5 months, approx. 7 years
Population: Clinical Database Population: All treated participants.
Measure: Number; unit: Participants
Arm/Group | Resistant/Intolerant Ph+ CML in CP | Newly Diagnosed and Untreated Ph+ CML in First CP
Number analyzed (Participants) | 33 | 25
Participants
  On-treatment deaths | 0 | 0
  Total Deaths | 1 | 3

ADVERSE EVENTS:
Time Frame: On treatment deaths were collected from FPFT up to 30 days after study drug discontinuation, for a maximum duration of 64.5 months (treatment duration ranged from 0.7 to 63.5 months). Deaths post treatment survival follow up were collected after the on- treatment period, up to approx. 7 years.
Description: Adverse Event: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment.
Groups:
- All Patients: All of the patients enrolled in the study.
Arm/Group | Resistant/Intolerant Ph+ CML in CP | Newly Diagnosed and Untreated Ph+ CML in First CP | All Patients
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/25 | 0/58
Serious Adverse Events (participants affected / at risk) | 11/33 | 4/25 | 15/58
Other Adverse Events (participants affected / at risk) | 33/33 | 25/25 | 58/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Resistant/Intolerant Ph+ CML in CP (N=33) | Newly Diagnosed and Untreated Ph+ CML in First CP (N=25) | All Patients (N=58)
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 1
Growth hormone deficiency (Endocrine disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
Haemorrhoids thrombosed (Gastrointestinal disorders) | 1 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 2 | 0 | 2
Hepatomegaly (Hepatobiliary disorders) | 1 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 1 | 2
Malaria (Infections and infestations) | 1 | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0 | 1
Tooth infection (Infections and infestations) | 1 | 0 | 1
Viral infection (Infections and infestations) | 1 | 1 | 2
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 1
Weight decreased (Investigations) | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1
Bone swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Jaw cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Facial paralysis (Nervous system disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 1 | 1
Syncope (Nervous system disorders) | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hyperaemia (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Resistant/Intolerant Ph+ CML in CP (N=33) | Newly Diagnosed and Untreated Ph+ CML in First CP (N=25) | All Patients (N=58)
Anaemia (Blood and lymphatic system disorders) | 4 | 3 | 7
Leukopenia (Blood and lymphatic system disorders) | 0 | 2 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3 | 4
Palpitations (Cardiac disorders) | 0 | 2 | 2
Gilbert's syndrome (Congenital, familial and genetic disorders) | 1 | 2 | 3
Ear pain (Ear and labyrinth disorders) | 1 | 2 | 3
Conjunctival haemorrhage (Eye disorders) | 0 | 2 | 2
Ocular hyperaemia (Eye disorders) | 1 | 3 | 4
Abdominal pain (Gastrointestinal disorders) | 3 | 6 | 9
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3 | 4
Constipation (Gastrointestinal disorders) | 1 | 2 | 3
Dental caries (Gastrointestinal disorders) | 3 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 7 | 4 | 11
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 2
Nausea (Gastrointestinal disorders) | 8 | 10 | 18
Odynophagia (Gastrointestinal disorders) | 0 | 2 | 2
Vomiting (Gastrointestinal disorders) | 7 | 8 | 15
Asthenia (General disorders) | 1 | 2 | 3
Fatigue (General disorders) | 0 | 6 | 6
Malaise (General disorders) | 2 | 1 | 3
Non-cardiac chest pain (General disorders) | 1 | 3 | 4
Pyrexia (General disorders) | 11 | 9 | 20
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 | 8 | 12
Seasonal allergy (Immune system disorders) | 2 | 1 | 3
Conjunctivitis (Infections and infestations) | 3 | 0 | 3
Cystitis (Infections and infestations) | 2 | 0 | 2
Ear infection (Infections and infestations) | 0 | 2 | 2
Gastroenteritis (Infections and infestations) | 0 | 6 | 6
Influenza (Infections and infestations) | 4 | 2 | 6
Nasopharyngitis (Infections and infestations) | 5 | 7 | 12
Otitis media acute (Infections and infestations) | 0 | 2 | 2
Parotitis (Infections and infestations) | 2 | 1 | 3
Pharyngitis (Infections and infestations) | 3 | 3 | 6
Rhinitis (Infections and infestations) | 4 | 4 | 8
Upper respiratory tract infection (Infections and infestations) | 10 | 7 | 17
Arthropod sting (Injury, poisoning and procedural complications) | 2 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 2
Joint injury (Injury, poisoning and procedural complications) | 2 | 0 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 2 | 2
Procedural pain (Injury, poisoning and procedural complications) | 3 | 1 | 4
Alanine aminotransferase increased (Investigations) | 10 | 11 | 21
Amylase increased (Investigations) | 3 | 0 | 3
Aspartate aminotransferase increased (Investigations) | 8 | 9 | 17
Blood bilirubin increased (Investigations) | 12 | 10 | 22
Blood cholesterol increased (Investigations) | 2 | 2 | 4
Blood creatine phosphokinase increased (Investigations) | 3 | 0 | 3
Blood creatinine increased (Investigations) | 0 | 2 | 2
Blood glucose increased (Investigations) | 2 | 1 | 3
Blood triglycerides increased (Investigations) | 0 | 2 | 2
Electrocardiogram QT prolonged (Investigations) | 5 | 1 | 6
Gamma-glutamyltransferase increased (Investigations) | 4 | 1 | 5
Lipase increased (Investigations) | 3 | 1 | 4
Neutrophil count decreased (Investigations) | 2 | 3 | 5
Platelet count decreased (Investigations) | 0 | 5 | 5
Weight decreased (Investigations) | 2 | 3 | 5
Weight increased (Investigations) | 1 | 3 | 4
Decreased appetite (Metabolism and nutrition disorders) | 5 | 1 | 6
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 4 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 4 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 7 | 16
Dizziness (Nervous system disorders) | 1 | 3 | 4
Headache (Nervous system disorders) | 13 | 14 | 27
Hypoaesthesia (Nervous system disorders) | 2 | 0 | 2
Paraesthesia (Nervous system disorders) | 2 | 2 | 4
Anxiety (Psychiatric disorders) | 1 | 2 | 3
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 3 | 4
Gynaecomastia (Reproductive system and breast disorders) | 2 | 2 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 7 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 9
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 5
Acne (Skin and subcutaneous tissue disorders) | 4 | 4 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 2 | 6
Dermatitis (Skin and subcutaneous tissue disorders) | 4 | 2 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 0 | 3
Erythema (Skin and subcutaneous tissue disorders) | 4 | 4 | 8
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Madarosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3 | 3
Rash (Skin and subcutaneous tissue disorders) | 7 | 11 | 18
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 3 | 8
Rash papular (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 1 | 4
Hypertension (Vascular disorders) | 3 | 2 | 5
Hypotension (Vascular disorders) | 3 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.